CLINICAL TRIAL: NCT02527109
Title: The Effect of Intra-anal Nifedipine, Used As Add-on to Conservative Therapy, on Pain in Patients With Anal Fissure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: RDD Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RDD 110
Record Dates: First submitted 2015-08-10; First posted 2015-08-18 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-06

CONDITIONS: Chronic Anal Fissure
MeSH Terms: interventions — Nifedipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Intra-anal placebo administered BID.
  Interventions: Drug: Nifedipine
- Nifedipine 12 mg/day (Experimental): Intra-anal Nifedipine 12 mg administered OD.
  Interventions: Drug: Nifedipine
- Nifedipine 24 mg/day (Experimental): Intra-anal Nifedipine 12 mg administered BID.
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Nifedipine

SUMMARY:
The objective of the study is to examine the effect of Nifedipine, applied intra-anally through our drug delivery device, on rectal pain severity in anal fissure patients that are being managed with conservative treatment.

DETAILED DESCRIPTION:
This is a randomized, double-blinded study. All patients in the study will be treated with the conservative standard of care for anal fissure. Study medication will be used as an add-on to conservative therapy, and will consist of 3 groups:

1. Treatment Group 1- 12 mg of Nifedipine to be self-administered twice daily.
2. Treatment Group 2- 12 mg of Nifedipine to be self-administered once daily in the morning hours and placebo to be self-administered in the evening.
3. Placebo Group - Placebo to be self-administered twice daily. Approximately 330 subjects will participate in this study. A screening visit will be used to determine subject suitability for inclusion in the trial. Within one week of the screening visit, subjects who meet all inclusion criteria and none of the exclusion criteria will receive either Nifedipine 12 mg X2 a day (BID) (24 mg/day total) or Nifedipine 12 mg X1/day to be administered in the morning hours and a matching placebo X1/day to be administered in the evening hours (12 mg/day total) or a matching placebo X2 a day (BID) (0 mg/day total) for a period of 8 weeks. During this period, 4 study visits (at 0, 2, 5, and 8 weeks) will take place. Study medication and placebo will be administered BID (in the morning and in the evening). In addition to receiving study medication, subjects will be maintained on a conservative standard treatment for Anal Fissure: sitz baths, high fiber diet, stool softeners and plenty of fluids.

Upon completion of the treatment cycle, patients will be contacted by phone (at weeks 10, 13 and 16) and will be questioned about recurrent symptoms e.g. pain or bleeding.

Patients that:

1. Were enrolled to one of the investigational groups ,and completed the 8 weeks treatment period or discontinued treatment because the investigator deemed them as healed AND
2. Experience symptoms of recurrence AND ARE
3. Willing to participate in an open label extension will receive Nifedipine 12 mg X2 a day (BID) for a period of 8 weeks. During this period, 4 study visits (at 0, 2, 5, and 8 weeks from the start of retreatment) will take place.

ELIGIBILITY:
Inclusion Criteria:

- Subjects meeting the following criteria will be eligible to participate in the trial:

1. Single anal fissure;
2. Signed written informed consent;
3. Male or female subjects 18 to 65 years of age inclusive;
4. Has chronic anal fissure defined as history of rectal pain at least three days a week for at least 6 weeks - or more AND at least one of the following:

   * Sentinel skin tag
   * Hypertrophied anal papilla
   * Exposure of the underlying internal anal sphincter
   * Anal cicatrisation
5. Visual analogue scale of average 24 hours rectal pain (VAS) of > 40 mm in screening visit
6. Capable of using the IVRS and able to adequately communicate comprehension of the IVRS questions to the investigator
7. If female, is non-lactating, has a negative urine pregnancy test result, and does not plan on becoming pregnant during the study, or not of childbearing potential (hysterectomy or tubal ligation at least 6 months prior to entry to the study or post-menopausal for 1 year); if of childbearing potential (including peri-menopausal women who have had a menstrual period within one year) must practice or be willing to continue to practice acceptable birth control from screening and until 1 week after the study medication has been discontinued.

Acceptable birth control includes :

* combined (estrogen and progestogen containing) hormonal contraception
* associated with inhibition of ovulation; oral OR intravaginal OR transdermal.
* progestogen-only hormonal contraception associated with inhibition of ovulation: oral OR injectable OR implantable.
* progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action
* intrauterine device (IUD)
* intrauterine hormone-releasing system ( IUS)
* bilateral tubal occlusion
* vasectomised partner
* sexual abstinence
* male or female condom with or without spermicide
* cap, diaphragm or sponge with spermicide

Exclusion Criteria:

* Subjects are excluded from participation in the study if any of the following criteria apply:

  1. Known allergy to Nifedipine
  2. Unwilling to stop all other concomitant topical preparations applied in and around the anus from screening through the end of the study
  3. Subfissure injection of botulinum toxin in the 3 months prior to screening.
  4. Fissure resulting from inflammatory bowel disease, venereal disease, perianal psoriasis, immunodeficiency syndrome
  5. Atypical fissure (occurs off the midline) in which secondary causes were not excluded.
  6. Deemed by the investigator as anal fissure for which surgery is indicated
  7. Anal abscess;
  8. Grade 4 hemorrhoids
  9. Fixed anal stenosis
  10. Active or past history of cardiovascular or cerebrovascular disease including but not limited to angina pectoris, myocardial infarction, transient ischemic attacks/stroke, arrhythmia or ecg changes that requires medical treatment or deemed by the investigator as clinically significant, moderate to severe congestive heart failure, or cardiac valve abnormalities;
  11. Type 1 diabetes mellitus
  12. Insulin treated type 2 diabetes mellitus
  13. Renal failure defined as a serum creatinine > 1.5 mg/dL (133 µmol/L) at screening
  14. Liver disease defined as Aspartate aminotransferase (AST) or alanine aminotransferase(ALT) >2 X upper limit of normal at screening
  15. Malignant disease within 3 years of screening
  16. Has uncontrolled hypertension (sitting blood pressure >160/95 mmHg at screening)
  17. Has hypotension (blood pressure lower than 90/60 mm Hg at screening)
  18. History of chronic gastrointestinal disease such as Crohn's disease or ulcerative colitis
  19. History of major rectal surgery
  20. History of HIV, Hepatitis B, Hepatitis C
  21. Has clinical laboratory test values (chemistry, hematology, or urinalysis) judged to be clinically significant by the investigator at screening;
  22. Has used, in the last two weeks, drugs that may affect blood coagulation, such as Aspirin at a dose higher than 500 mg/day, Warfarin, Sintrom, Enoxaparin, Nadroparin, Heparin, Clopidogrel, Ticlopidine Rivaroxaban, Apixaban, Edoxaban
  23. Is treated with drugs that may affect the anal sphincter:

      1. Calcium channel blockers such as Nifedipine, Diltiazem or Verapamil
      2. Nitroglycerin or nitrates
  24. Has, upon physical examination, a rectal deformation or signs of rectal disease such as fistula, infection or space occupying lesion;
  25. Participated in a clinical study in the last 30 days prior to screening.
  26. Is an immediate family member of personnel directly affiliated with the study at the investigative site, or is personally directly affiliated with the study at the investigative site; or is employed or related to the Sponsor, CRO or investigator;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2016-05; Primary Completion 2018-06-15 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Rectal pain and measured by VAS | measured at day 56

SECONDARY OUTCOMES:
Healing of anal fissure | day 56
  Healing is defined by lack of pain AND evidence of epithelization in a physical examination

CONTACTS AND LOCATIONS:
Locations (24):
- Bulgaria (7):
  - UMHAT "Sveti Georgi", Internal Consulting Department, Plovdiv
  - "Multiprofile Hospital for Active Treatment - Doverie" AD, Clinic of Gastroenterology, Sofia
  - II MHAT, Internal Clinic, Department of Gastroenterology, Sofia
  - MC Health BG EOOD, Sofia
  - Multiprofile Hospital for Active Treatment Lulin, Sofia
  - MC "New rehabilitation centre'' EOOD, Stara Zagora
  - "Multiprofile Regional Hospital for Active Treatment - Dr. St. Cherkezov" AD Department of Gastroenterology, Veliko Tarnovo
- Moldova (3):
  - IMSP Spitalul Clinic Municipal Nr 1, Chisinau
  - IMSP Spitalul Clinic Municipal Nr 3 "Sfanta Treime", Chisinau
  - IMSP Spitalul Clinic Republican, Chisinau
- Poland (4):
  - Med-Gastr Centrum Medyczne, Lodz
  - Ambulatorium Medyczne Medical Hair & Esthetic, Lublin
  - Centrum Innowacyjnych Terapii Sp. z o.o. Oddział w Piasecznie, Piaseczno
  - NZOZ Specjalistyczne Centrum Medyczne Flebo, Wołomin
- Romania (10):
  - Pelican Impex SRL, Oradea, Jud. Bihor
  - Institutul Regional de Gastroenterologie si Hepatologie "Prof. Dr. Octavian Fodor", Cluj-Napoca, Jud. Cluj
  - IRGH, Cluj-Napoca, Jud. Cluj
  - Tvm Med Serv Srl, Cluj-Napoca, Jud. Cluj
  - SC Schnelbach Medical Care SRL, Ploieşti, Jud. Prahova
  - Spit. Clinic Judetean de Urgenta "Sf. Apostol Andrei" Constanta, Constanța, Judet Constanta
  - Dacmed SRL, Ploieşti, Prahova
  - Centrul Medical de Diagnostic si Tratament Ambulator Neomed SRL, Brasov
  - Institutul Clinic Fundeni, Bucharest
  - Centrul Medical Sfanta Vineri SRL, Bucharest